CLINICAL TRIAL: NCT06723743
Title: Transcutaneous Auricular Vagus Nerve Stimulation Effects on Attention and Working Memory: A Pilot Study
Brief Title: Transcutaneous Vagus Nerve Stimulation for Attention and Memory
Acronym: taVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ricardo Jorge, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-56468
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury (TBI) Patients
Keywords: vagus nerve stimulation; attention; brain stimulation; PTSD; depression
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Depression | interventions — Whole-Body Irradiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- taVNS active stimulation (Active Comparator): Participants will receive transcutaneous auricular vagus nerve stimulation (taVNS) using electrodes placed on the left ear. A low-level electrical current will be delivered to stimulate the vagus nerve. This stimulation is designed to activate brain areas involved in attention and memory.
  Interventions: Other: Transcutaneous vagus nerve stimulation for attention in veterans with TBI; Device: Soterix Medical Vagus Nerve Stimulation mini-CT
- Sham (Placebo) taVNS (Sham Comparator): Participants will undergo sham stimulation, where electrodes are placed on the left ear to mimic the experience of active taVNS. However, no electrical current will be delivered to the vagus nerve. This sham condition enables a direct comparison with active taVNS, ensuring that any observed changes in working memory and attention can be attributed to the taVNS intervention.
  Interventions: Other: Transcutaneous vagus nerve stimulation for attention in veterans with TBI; Device: Soterix Medical Vagus Nerve Stimulation mini-CT

INTERVENTIONS:
Other: Transcutaneous vagus nerve stimulation for attention in veterans with TBI — taVNS does not require surgery or medication, offering a safe and accessible treatment option. Each participant undergoes both an active taVNS session and a sham (placebo) session. Sham stimulation mimics the sensory experience of taVNS but does not deliver electrical currents to the vagus nerve, ensuring blinding and providing robust comparisons. The study is completed in a single visit lasting 2.5 to 3 hours, minimizing participant burden.
Device: Soterix Medical Vagus Nerve Stimulation mini-CT — Soterix Medical min-CT VNS device is used for non-invasive stimulation procedures and trials. It has blinding features such as single-blind for this study in which patients will either receive active or shame taVNS.

SUMMARY:
This clinical trial aims to evaluate whether transcutaneous auricular vagus nerve stimulation (taVNS), a non-invasive brain stimulation method, can improve attention and memory in veterans with traumatic brain injury (TBI) and depression and/or posttraumatic stress disorder (PTSD). The study seeks to answer two main questions:

1. Can active taVNS improve attention and memory compared to sham (placebo) stimulation?
2. Does taVNS affect heart rate variability (HRV)?

taVNS delivers a gentle electrical current to the vagus nerve through electrodes placed on the ear, targeting brain areas involved in attention and memory without requiring surgery.

This study uses a crossover design, meaning all participants will experience two sessions: one with active taVNS and one with sham stimulation. The sham session feels similar but does not deliver actual stimulation, allowing researchers to compare the two and understand taVNS's effects on the brain.

In a single visit, participants will:

* Complete eligibility screening (questionnaires and vital signs).
* Undergo two sessions (one active and one sham), randomly assigned.
* Perform attention tasks before and after each session.
* Have their heart rate monitored during the sessions.

The findings will help determine whether taVNS could be an effective treatment for improving attention and memory in veterans with TBI.

DETAILED DESCRIPTION:
Attention and memory problems are common in veterans with traumatic brain injuries (TBI), particularly when accompanied by depression and/or posttraumatic stress disorder (PTSD). Current treatments for these issues often have limited effectiveness or unwanted side effects. Transcutaneous auricular vagus nerve stimulation (taVNS) is a non-invasive technique that uses gentle electrical impulses delivered through electrodes placed on the ear. This stimulation targets the vagus nerve, which plays a key role in regulating brain areas involved in attention and memory. By enhancing the activity of these brain regions, taVNS shows potential as a novel treatment option for improving cognitive functions like attention and memory.

In this study, researchers aim to determine whether taVNS can enhance attention and memory in veterans with TBI. Participants will complete a single study visit lasting 2.5 to 3 hours. The visit includes two taVNS sessions, one active and one sham (placebo), to compare their effects. Sham stimulation mimics the sensation of taVNS but does not deliver electrical current to the vagus nerve. This design allows researchers to isolate the specific effects of taVNS.

Procedures:

1. Screening (40 minutes):

   Participants will begin by completing questionnaires about their medical history, memory concerns, alcohol and substance use, mood, and demographics. Vital signs (heart rate, blood pressure, and temperature) will also be measured to confirm eligibility.
2. Session 1 (approximately 40 minutes):

   Participants will complete a computer-based attention task that involves responding to specific visual cues on a screen. This task takes about 10 minutes. taVNS will then be delivered using electrodes placed on the left ear. For this session, participants will either receive active stimulation or sham stimulation, randomly assigned. The stimulation lasts 20 minutes. After the stimulation, participants will repeat the attention task to assess changes in performance.
3. Break:

   Participants will have a short break between sessions, during which they can rest or engage in light activities.
4. Session 2 (approximately 40 minutes):

The same sequence of procedures will be repeated, but participants will receive the alternate type of stimulation (active or sham) in this session. The order of active and sham stimulation is randomly assigned, and participants will not know which session is delivered first.

Throughout both sessions, participants' heart rate variability (HRV) will be monitored using a lightweight chest device. HRV provides insights into how the body responds to stimulation and helps evaluate taVNS's physiological effects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-64
* Right-handedness
* Veterans with a history of deployment to Operation Iraqi Freedom (OIF), Operation Enduring Freedom (OEF), Operation New Dawn (OND) or other post 9/11 war on terrorism
* History of PTSD and/or depression
* Military related mild traumatic brain injury
* If taking psychotropic medication, demonstrate stability for 3 months
* If taking stimulants, washout period of 12 hours

Exclusion Criteria:

* History of neurological, cardiovascular, or pulmonary disease
* Cardiac arrhythmia (all types)
* Active suicidal ideation
* Visible wounds on skin of the left ear
* Medical implants such as cardiac defibrillators, pacemakers, or deep brain stimulators
* Pregnancy
* Completed taVNS in the past 4 weeks
* Current substance use disorder (exception: mild cannabis use disorder allowed)
* Current moderate or severe alcohol use disorder
* Major cognitive disorder

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Attention and working memory | One day, one visit
  Aim 1:
  To evaluate the effects of transcutaneous auricular vagus nerve stimulation (taVNS) on sustained attention and working memory. Attention and memory performance will be assessed using the Gradual Onset Continuous Performance Task (gradCPT), a validated computerized test that measures the ability to sustain attention and respond selectively to relevant stimuli. This cognitive test measures sustained attention and inhibitory control. During the test, subjects view a continuous stream of gradually fading images of cities and mountains on a computer screen. They are instructed to press the space bar when they see a city (target stimulus) and withhold responses when they see a mountain (non-target stimulus). Key performance metrics which collectively assess attention and working memory in this test include mean reaction time (response speed), omission errors (failure to respond to targets), and commission errors (responses to non-targets).

SECONDARY OUTCOMES:
Heart-rate variability | One day, one visit
  Aim 2: To investigate the effects of taVNS on heart rate variability (HRV), an indicator of autonomic nervous system activity. HRV will be measured in milliseconds using a lightweight, wearable chest device capable of capturing continuous heart rate data. Key HRV metrics, including standard deviation of NN intervals (SDNN) and root mean square of successive differences (RMSSD), will be analyzed before, during, and after active and sham taVNS sessions to assess physiological responses to stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is an exploratory, feasibility trial designed to assess the potential effects of transcutaneous auricular vagus nerve stimulation (taVNS). As a pilot study, the primary goal is to evaluate the intervention's feasibility and gather preliminary data, rather than generate findings intended for broader generalization. To protect participant privacy and confidentiality, all data will be reported in aggregate form without identifying individual participants, in accordance with ethical guidelines and institutional policies.

REFERENCES:
- [Background] Stefan H, Kreiselmeyer G, Kerling F, Kurzbuch K, Rauch C, Heers M, Kasper BS, Hammen T, Rzonsa M, Pauli E, Ellrich J, Graf W, Hopfengartner R. Transcutaneous vagus nerve stimulation (t-VNS) in pharmacoresistant epilepsies: a proof of concept trial. Epilepsia. 2012 Jul;53(7):e115-8. doi: 10.1111/j.1528-1167.2012.03492.x. Epub 2012 May 3. PMID 22554199
- [Background] Sun JB, Cheng C, Tian QQ, Yuan H, Yang XJ, Deng H, Guo XY, Cui YP, Zhang MK, Yin ZX, Wang C, Qin W. Transcutaneous Auricular Vagus Nerve Stimulation Improves Spatial Working Memory in Healthy Young Adults. Front Neurosci. 2021 Dec 23;15:790793. doi: 10.3389/fnins.2021.790793. eCollection 2021. PMID 35002607
- [Background] Schein J, Adler LA, Childress A, Gagnon-Sanschagrin P, Davidson M, Kinkead F, Cloutier M, Guerin A, Lefebvre P. Economic burden of attention-deficit/hyperactivity disorder among adults in the United States: a societal perspective. J Manag Care Spec Pharm. 2022 Feb;28(2):168-179. doi: 10.18553/jmcp.2021.21290. Epub 2021 Nov 22. PMID 34806909
- [Background] Ruffoli R, Giorgi FS, Pizzanelli C, Murri L, Paparelli A, Fornai F. The chemical neuroanatomy of vagus nerve stimulation. J Chem Neuroanat. 2011 Dec;42(4):288-96. doi: 10.1016/j.jchemneu.2010.12.002. Epub 2010 Dec 16. PMID 21167932
- [Background] Perugi G, De Rosa U, Barbuti M. What value do norepinephrine/dopamine dual reuptake inhibitors have to the current treatment of adult attention deficit hyperactivity disorder (ADHD) treatment armamentarium? Expert Opin Pharmacother. 2022 Dec;23(18):1975-1978. doi: 10.1080/14656566.2022.2148830. Epub 2022 Nov 16. No abstract available. PMID 36384367
- [Background] Nasiri, E., Khalilzad, M., Hakimzadeh, Z. et al. A comprehensive review of attention tests: can we assess what we exactly do not understand?. Egypt J Neurol Psychiatry Neurosurg 59, 26 (2023). https://doi.org/10.1186/s41983-023-00628-4
- [Background] Konjusha A, Colzato L, Muckschel M, Beste C. Auricular Transcutaneous Vagus Nerve Stimulation Diminishes Alpha-Band-Related Inhibitory Gating Processes During Conflict Monitoring in Frontal Cortices. Int J Neuropsychopharmacol. 2022 Jun 21;25(6):457-467. doi: 10.1093/ijnp/pyac013. PMID 35137108
- [Background] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Background] Geng D, Liu X, Wang Y, Wang J. The effect of transcutaneous auricular vagus nerve stimulation on HRV in healthy young people. PLoS One. 2022 Feb 10;17(2):e0263833. doi: 10.1371/journal.pone.0263833. eCollection 2022. PMID 35143576
- [Background] Foley JO, and DuBois FS (1937). Quantitative studies of the vagus nerve in the cat. J Comp Neurol 67, 49-67.
- [Background] Eriksson J, Vogel EK, Lansner A, Bergstrom F, Nyberg L. Neurocognitive Architecture of Working Memory. Neuron. 2015 Oct 7;88(1):33-46. doi: 10.1016/j.neuron.2015.09.020. PMID 26447571
- [Background] Cowan N. The many faces of working memory and short-term storage. Psychon Bull Rev. 2017 Aug;24(4):1158-1170. doi: 10.3758/s13423-016-1191-6. PMID 27896630
- [Background] Constantinidis C, Klingberg T. The neuroscience of working memory capacity and training. Nat Rev Neurosci. 2016 Jul;17(7):438-49. doi: 10.1038/nrn.2016.43. Epub 2016 May 26. PMID 27225070
- [Background] Badran BW, Yu AB, Adair D, Mappin G, DeVries WH, Jenkins DD, George MS, Bikson M. Laboratory Administration of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS): Technique, Targeting, and Considerations. J Vis Exp. 2019 Jan 7;(143):10.3791/58984. doi: 10.3791/58984. PMID 30663712
- [Background] Arakaki X, Arechavala RJ, Choy EH, Bautista J, Bliss B, Molloy C, Wu DA, Shimojo S, Jiang Y, Kleinman MT, Kloner RA. The connection between heart rate variability (HRV), neurological health, and cognition: A literature review. Front Neurosci. 2023 Mar 1;17:1055445. doi: 10.3389/fnins.2023.1055445. eCollection 2023. PMID 36937689
- [Background] Aniwattanapong D, List JJ, Ramakrishnan N, Bhatti GS, Jorge R. Effect of Vagus Nerve Stimulation on Attention and Working Memory in Neuropsychiatric Disorders: A Systematic Review. Neuromodulation. 2022 Apr;25(3):343-355. doi: 10.1016/j.neurom.2021.11.009. Epub 2022 Jan 26. PMID 35088719